CLINICAL TRIAL: NCT04872465
Title: Efficacy of Bilateral Dorsolateral Prefrontal Theta-burst Stimulation in Elderly Refractory Depression: a Randomized Sham-controlled Study
Brief Title: TBS Over DLPFC in Elderly Refractory Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Che-Sheng Chu, Department of Psychiatry, MD, attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kaohsiung VGHKS
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): We initially used cTBS (continuous TBS) over right DLPFC with 120-s train of uninterrupted bursts (1800 pulses) in each session per day. After that, we continuous use iTBS (intermittent TBS, iTBS) over left DLPFC with 2-s train of bursts was repeated every 10 s for a total of 570 s (1800 pulses).
  Interventions: Device: TBS
- Sham Comparator (Placebo Comparator): Participants will receive sham (placebo) TBS treatment the same as experimental group
  Interventions: Device: sham

INTERVENTIONS:
Device: TBS — We initially used cTBS (continuous TBS) over right DLPFC with 120-s train of uninterrupted bursts (1800 pulses) in each session per day. After that, we continuous use iTBS (intermittent TBS, iTBS) over left DLPFC with 2-s train of bursts was repeated every 10 s for a total of 570 s (1800 pulses).
  Arms: Experimental
Device: sham — Participants will receive sham (placebo) TBS treatment the same as experimental group
  Arms: Sham Comparator

SUMMARY:
The study aim to examine the effect of Thea-burst stimulation over bilateral dorsolateral prefrontal cortex (DLPFC) among patients with LLD on mood condition and relevant biomarkers.

DETAILED DESCRIPTION:
Thea-burst stimulation (TBS) is a novel form of rTMS, providing greater modulation effect on neural activity. So far, no study was conducted to use TBS as treatment in LLD. Therefore, we aim to examine the effect of TBS over bilateral dorsolateral prefrontal cortex (DLPFC) among patients with LLD on mood condition and relevant biomarkers. The study used a two-arm, parallel, double-blind, randomized, and sham-controlled design. We plan to enroll sixty patients with LLD, thirty for active intervention and thirty for sham-controlled group. An Magstim Rapid2 stimulator with eight-figure coil was used for stimulation. Location of brain area are based on bilateral DLPFC. 3-pulse 50-Hz bursts was given every 200ms (at 5 Hz) and an intensity of 80% active motor threshold was settled. We initially used cTBS (continuous TBS) over right DLPFC with 120-s train of uninterrupted bursts (1800 pulses) in each session per day. After that, we continuous use iTBS (intermittent TBS, iTBS) over left DLPFC with 2-s train of bursts was repeated every 10 s for a total of 570 s (1800 pulses). Each patient received daily stimulation for two weeks with total ten sessions. The primary outcomes were change of depression severity including response and remission rate. Secondary outcome were biomarkers related to depression. Assessments were administered at baseline, immediately after 5 and 10 sessions of stimulation, and 3 months after the completion of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 85 years
* Major depression disorder
* Under a stable dose of all psychotropic medication during the stimulation period.

Exclusion Criteria

* Having any current psychiatric comorbidity or history of substance dependence.
* Having active suicidal ideation currently.
* Having severe physical illness, recent and/or current unstable medical disorders.
* Having history of cancer or chemotherapy.
* Dementia or MMSE<24.
* Having TMS contraindicated (seizure disorder, history of seizures, metal in the head, pacemakers, history of craniotomy)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale, HAM-D | Change from baseline after 1, 2 weeks and three months
  The Ham-D is the most widely used clinician-administered depression assessment scale. The original version contains 17 items pertaining to symptoms of depression experienced over the past week. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.

SECONDARY OUTCOMES:
Beck depression inventory, BDI-II | Change from baseline after 1, 2 weeks and three months
  The BDI-II was a 1996 revision of the BDI. Participants were asked to rate how they have been feeling for the past two weeks. BDI-II also contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used as follows: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
Beck anxiety inventory, BAI | Change from baseline after 1, 2 weeks and three months
  The BAI, created by Aaron T. Beck and other colleagues, is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults. The BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms. The standardized cutoffs are as follows: 0-7: minimal anxiety; 8-15: mild anxiety; 16-25: moderate anxiety; 26-63: severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Che-Sheng Chu, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Department of Psychiatry, Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No